CLINICAL TRIAL: NCT04292886
Title: Hormone Replacement Versus Tamoxifen Combined Of Hormone Replacement in Women With a Thin Endometrium Undergoing Frozen-thawed Embryo Transfer
Brief Title: Thin Endometrium Undergoing Frozen-thawed Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Qingqing Shi, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NanjingU
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Thin Endometrium
Keywords: thin endometrium
MeSH Terms: interventions — Tamoxifen; femoston; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- thin endometrium ,treatment,Tamoxifen (Active Comparator): From the 2nd day of the menstrual cycle, the patient took tamoxifen and femoston
  Interventions: Drug: Tamoxifen and femoston
- thin endometrium ,treatment,Vitamin C (Placebo Comparator): From the 2nd day of the menstrual cycle, the patient took Vitamin C and femoston
  Interventions: Drug: Vitamin C and femoston

INTERVENTIONS:
Drug: Tamoxifen and femoston — oral
  Arms: thin endometrium ,treatment,Tamoxifen
Drug: Vitamin C and femoston — Vitamin C and femoston
  Arms: thin endometrium ,treatment,Vitamin C

SUMMARY:
The endometrium is essential for embryo implantation. The clinical pregnancy rate and live birth rate of patients with thin endometrium are significantly lower than those of normal endometrium. Previous studies have shown that tamoxifen has advantages for improving endometrial thickness. However, there is still a lack of evidence from randomized clinical trials comparing the efficacy between hormone replacement and Tamoxifen combined Of hormone replacement.This is a prospective, randomized placebo-controlled, double-blind clinical trial that includes 120 patients younger than 38 years old with a thin endometrium preparing for frozen embryo transfer. Participants will be randomly assigned (1: 1) into two parallel groups: estrogen replacement and tamoxifen combined with estrogen replacement.Frozen embryo resuscitation transfer cycle for thin endometrium patients。This is the first randomized controlled trial to comparing estrogen and estrogen combined with tamoxifen for endometrial improvement，The results of this study will provide evidence for the efficacy of the strategy of frozen embryo transfer cycle for thin endometrium patients.

ELIGIBILITY:
Inclusion Criteria:

1) Younger than 38 years old, basal serum level of follicle stimulating hormone <10 IU / L; (2) Endometrium is less than 8mm in at least 2 cycles: superovulation cycle / natural cycle / estrogen replacement therapy / ovarian stimulation cycle; (3) at least 1 high quality frozen embryo; (4) There are no comorbidities that clearly affect pregnancy, such as adenomyosis, endometriosis, and intrauterine adhesions;

Exclusion Criteria:

1. abnormal karyotype;
2. Accompanying other diseases of the uterus: uterine muscular wall myomas that affect the uterine cavity shape, more severe adenomyosis, severe endometriosis, congenital uterine malformations, endometrial tuberculosis, etc .;
3. Contraindications to hormone replacement therapy;
4. Participating in other clinical research;
5. History of previous fundus diseases;

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness | within the 15 days (plus or minus 5 days) after oral drugs
  Endometrial thickness were record using transvaginal ultrasound scan.

CONTACTS AND LOCATIONS:
Overall Officials: Haixiang Sun, Ph.D, Principal Investigator — Nanjing University Medical School Affiliated Nanjing Drum Tower Hospital
Locations (1):
- Nanjing University Medical School Affiliated Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China